CLINICAL TRIAL: NCT06176534
Title: Combination Followed by Maintenance Chemotherapy Versus CDK4/6 Inhibitor Combined With Endocrine Therapy for HR Low/HER2-negative Advanced Breast Cancer: a Prospective, Randomized, Open-label Phase Ⅱ Clinical Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Min Yan, MD, Chief Physician, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HNCH-MBC013
Record Dates: First submitted 2023-12-09; First posted 2023-12-19 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Advanced Breast Cancer; Treatment; HR Low/HER2 Negative
MeSH Terms: interventions — Vinorelbine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): nab-paclitaxel 130mg/m2，day 1 and day 8 Capecitabine 2000mg/m2，from day1 to DAY 14 Vinorelbine 25mg/m2，day 1 and day 8
  Interventions: Drug: Experimental: chemotheyapy
- B (Active Comparator): palbociclib/Dalpiciclib Letrozole/Anastrozole/fulvestrant
  Interventions: Drug: Active Comparator: endocrine therapy

INTERVENTIONS:
Drug: Experimental: chemotheyapy — nab-paclitaxel 130mg/m2，day 1 and day 8 + Capecitabine 2000mg/m2, followed by nab-paclitaxel 130mg/m2，day 1 and day 8 or Capecitabine from day1 to DAY 14 Vinorelbine 25mg/m2，day 1 and day 8 + Capecitabine 2000mg/m2，from day1 to DAY 14
  Other Names: Vinorelbine 25mg/m2，day 1 and day 8 + Capecitabine 2000mg/m2，from day1 to DAY 14
  Arms: A
Drug: Active Comparator: endocrine therapy — palbociclib 125mg per day for 21days Dalpiciclib 150mg per day for 21days Letrozole 2.5mg per day Anastrozole 1mg per day fulvestrant 500mg per 28 days
  Arms: B

SUMMARY:
To observe the differences in the efficacy of Combination followed by maintenance chemotherapy versus CDK4/6 inhibitor combined with endocrine therapy in HR low expression /HER2 negative advanced breast cancer, and to provide new evidence for the best treatment of HR low expression /HER2 negative advanced breast cancer, and to explore the efficacy and safety of combined/maintenance chemotherapy.

DETAILED DESCRIPTION:
To observe the differences in the efficacy of Combination followed by maintenance chemotherapy versus CDK4/6 inhibitor combined with endocrine therapy in HR low expression /HER2 negative advanced breast cancer, and to provide new evidence for the best treatment of HR low expression /HER2 negative advanced breast cancer, and to explore the efficacy and safety of combined/maintenance chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years old; Invasive breast cancer with metastatic disease confirmed by histological or cytological examination; Patients without pathologically or cytologically confirmed metastatic disease should have clear evidence of metastasis by physical examination or radiological studies;
2. The most recent pathological report of biopsy confirmed HR low expression and HER2 negative.

   1. HR low expression was defined as 1-50% ER expression by immunohistochemistry (IHC); Or ER<1% and PR≥1%; Patients with ER expression of 1-10% or ER-/ PR-positive patients were eligible for inclusion after careful evaluation by the investigator, and those with a small tumor burden and candidates for endocrine therapy were eligible.
   2. HER2-negative definition: IHC 0 or 1+; If the IHC was 2+, it was confirmed negative by fluorescence in situ hybridization (FISH).
3. at least one measurable lesion;
4. No previous salvage chemotherapy for metastatic disease was required, and first-line endocrine therapy was allowed;
5. no previous CDK4/6 inhibitor; For adjuvant CDK4/6i treatment, recurrence and metastasis were required more than 1 year after drug withdrawal.
6. Eastern Cooperative Oncology Group performance status (ECOG PS) 0-1, life expectancy is more than 12 weeks;
7. Adequate function of major organs.
8. All adverse events recovered to grade 1 or less before enrollment (NCI CTCAE version 5.0);
9. patients without major organ dysfunction and heart disease;
10. Women and men of childbearing potential must agree to use appropriate contraception before and during study participation.

Exclusion Criteria:

1. symptomatic, uncontrolled brain or leptomeningeal metastases; Patients who had received previous systemic radical treatment for brain metastases (radiotherapy or surgery), if stable disease had been maintained for at least 1 month as confirmed by imaging, and if systemic hormone therapy (dose 10mg/ day prednisone or other effective hormones) for more than 2 weeks without clinical symptoms.
2. patients received radiotherapy, chemotherapy, major surgery, targeted therapy or immunotherapy within 2 weeks before enrollment; Patients received endocrine therapy within 1 week before enrollment. Chemotherapy with nitrosourea or mitomycin was administered within 6 weeks before enrollment.
3. participated in other clinical trials of new drugs within 4 weeks before enrollment;
4. there can not be controlled by drainage or pneumatic methods third space effusion;
5. patients with other malignant tumors within the past 3 years, excluding radical cervical carcinoma in situ, skin basal cell carcinoma or skin squamous cell carcinoma;
6. suffering from serious or uncontrolled diseases, including but not limited to: 1) active viral infection, such as HIV or HBV active (HbsAg positive and HBV-DNA≥103, hepatitis C antibody positive); 2) history of severe cardiovascular disease: uncontrolled hypertension; Myocardial infarction, unstable arrhythmia, congestive heart failure, pericarditis, myocarditis, etc. Patients with NYHA class ⅲ-ⅳ cardiac dysfunction, or left ventricular ejection fraction (LVEF) 50% by echocardiography; 3) severe infection (e.g., intravenous antibiotic, antifungal, or antiviral therapy according to clinical practice) within 4 weeks prior to the first dose or unexplained fever during screening/before the first dose; 38.3°C (fever due to cancer, as judged by the investigator, was eligible);
7. patients with a history of psychotropic drug abuse and unable to abstain or with mental disorders; Or accompanied by swallowing and absorption dysfunction;
8. patients with other concomitant diseases that seriously endanger the safety of patients or affect the completion of the study according to the judgment of the investigators;
9. patients with known history of allergy to the components of this regimen; A history of immunodeficiency, including testing positive for HIV, HCV or other acquired or congenital immunodeficiency disorders, or a history of organ transplantation;
10. pregnant or lactating women;
11. Patients deemed unsuitable for inclusion by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
ORR by investigator using RECIST Guideline (Version 1.1) | 6 weeks
  ORR was defined as percentage of participants with best (confirmed) overall response (BOR) of either CR or PR assessed by the investigator according to RECIST version 1.1

SECONDARY OUTCOMES:
PFS | up to 1.5 years
  PFS was defined as the time from first dose to first documented disease progression (PD) or death from any cause, whichever occurred first
Adverse events | up to 1.5 years
  Proportion of participants experienced adverse events during the study period
OS | up to 3 years
  OS was defined as the time from first dose to death for any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Breast Cancer Center, The Affiliated Cancer Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No